CLINICAL TRIAL: NCT04581122
Title: Zhongshan Hospital
Brief Title: A Multiple-center Study on the Effect of Different Ways of Lymph Node Dissection on the Prognosis of Ground Glass Nodules Smaller Than 3cm and With More Than 50% Solid Components
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2020-164R
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Progression
MeSH Terms: conditions — Disease Progression | interventions — Lymph Node Excision

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective lymphadenectomy (Experimental)
  Interventions: Procedure: Lymphadenectomy
- Systematic lymph node dissection (No Intervention)

INTERVENTIONS:
Procedure: Lymphadenectomy — Patients with ground glass nodules smaller than 3cm and with more than 50%solid components would randomly assigned to selective lymphadenectomy group or systematic lymph node dissection group
  Arms: Selective lymphadenectomy

SUMMARY:
A multiple-center study on the effect of different ways of lymph node dissection on the prognosis of less than 3cm ground glass nodules with more than solid components

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years;
2. GGO is diagnosed by lung CT and failure to subside after 3 months (the patient having been re-examined by thin-section CT);
3. The maximum diameter of the GGO is smaller than 3cm;
4. The maximum diameter of the solid component in the GGO is more than 50%;
5. The patient is able to undergo the lobectomy
6. The patient is able to understand and comply with the study and has provided written informed consent.

Exclusion Criteria:

-

Patients meeting any of the following criteria are not eligible for this trial:

1. Patients with a history of using immunosuppressive or hormonal drugs;
2. Patients receiving radiotherapy or chemotherapy;
3. Patients who fail to comply with our follow-up strategy;
4. Other situations that are not in conformity with the standards and requirements of this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 5 years
  five year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wei, Study Director — Fudan University
Locations (1):
- Jiang Wei, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided